CLINICAL TRIAL: NCT04818099
Title: A Multicenter, Randomized, Double-blind, Controlled Clinical Trial of Votioxetine in the Treatment of Depression After Radiotherapy for Head and Neck Cancer
Brief Title: Vortioxetine in the Treatment of Depression Associated With Head and Neck Cancers Undergoing Radiotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Brain Hospital Affiliated to Guangzhou Medical University (Unknown)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200813
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Radiation Injuries
Keywords: Vortioxetine; Depression; Cognitive function; Head and Neck Cancers
MeSH Terms: conditions — Radiation Injuries; Depression; Head and Neck Neoplasms | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine supportive psychotherapy and votioxetine (Experimental): On the basis of general psychotherapy, cognitive behavior therapy and supportive psychotherapy, the patients were given votioxetine 10mg/tablet, one tablet each time, once a day, for 2 months.
  Interventions: Drug: Vortioxetine 10 mg
- routine supportive psychotherapy and control (Placebo Comparator): On the basis of general psychotherapy, cognitive behavior therapy and supportive psychotherapy, the patients were given placebo, one tablet each time, once a day, for 2 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vortioxetine 10 mg — Vortioxetine will be used with a dosage of 10mg once a day, for 2 months.
  Arms: routine supportive psychotherapy and votioxetine
Other: Placebo — Placebo will be used with a dosage of one tablet once a day for 2 months.
  Arms: routine supportive psychotherapy and control

SUMMARY:
The purpose of this study is to evaluate the effects of vortioxetine, once daily (QD), on mood disorders and cognitive dysfunction in patients with head and neck cancers undergoing radiotherapy.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the fifth most common cancer in the world, especially in South China. The incidence of depression and anxiety in HNC patients after radiotherapy is as high as 12% - 45% due to appearance changes, decreased swallowing function, dry mouth, pain and other discomfort. At the same time, radiotherapy, as mainstay of therapy for HNC, also causes different degrees of damage to the brain around the tumor, leading to secondary cognitive dysfunction. Depression, anxiety and cognitive impairment seriously affect the quality of life of HNC patients after radiotherapy. Recent studies have found that votioxetine has multimodal pharmacodynamic activity, which can not only improve symptoms of depression, but also significantly improve the cognitive function of patients. In this study, investigators will discuss the therapeutic effect of vortioxetine on the depression after radiotherapy in HNC patients through a multi-center, randomized and double-blind comparative clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* (1) Received radiation therapy due to head and neck cancer.
* (2) The patient have depression symptoms (PHQ-9 score ≥ 8) and meet the ICD-10 (version 2019) diagnostic criteria.
* (3) Age>/= 18 years and age</=65.
* (4) Estimated life expectancy ≥ 12 months.
* (5) Constant caregivers who well understand and have willingness to sign a written informed consent document.

Exclusion Criteria:

* (1) The researcher believe that the subjects have the tendency of suicide, self mutilation or the score of "suicide concept" in item 10 of MADRS was ≥5, or they had committed suicide, self mutilation within 6 months before enrollment;
* (2) History of depressive disorder before radiotherapy for head and neck tumors;
* (3) History of other serious mental disorders, such as generalized anxiety disorder, drug and alcohol abuse, etc;
* (4) History of central nervous diseases such as Alzheimer's disease, Parkinson's disease, Stroke, uncontrolled epilepsy, etc., which lead to emotional and cognitive impairment and other serious and uncontrolled systemic diseases (such as cardiopulmonary insufficiency, etc.);
* (5) Baseline Mini Mental State Examination (MMSE) score ≤ 23 points (University or above), MMSE ≤ 22 points (middle school), MMSE ≤ 20 points (primary school), MMSE ≤ 17 points (illiteracy);
* (6) The subject with brain metastasis;
* (7) Hematological examination of subject: White blood cell count < 3.5×10^9/L, Platelet count < 100×10^9/L, Hemoglobin < 110g/L, Abnormal range of coagulation function like fibrinogen < 1.5g/L, or other coagulation abnormalities with clinical significance；
* (8) Blood biochemical examination of patients: Total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2.0 x upper limit of normal value, Creatinine > 1.5x upper limit of normal value, Blood sodium < 130mmol/L;
* (9) The subject has a history of severe drug allergy or is known to be allergic to any excipient of the test drug;
* (10) The subjects who could not effectively complete the neuropsychological test during the follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 8 in the MADRS Total Score | Baseline to Week 8
  MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms.

SECONDARY OUTCOMES:
Change From Baseline to Week 8 in the Digit Symbol Substitution Test (DSST) | Baseline to Week 8
  The DSST assesses relative contributions of speed, memory, executive function and visual scanning. Higher scores-correct number of symbols reflects greater objective cognitive functioning.
Change from baseline to 8 weeks in Rey Auditory Verbal Learning Test (RAVLT) | Baseline to Week 8
  The purpose of the RAVLT is to assess verbal learning and memory. Specifically, it assesses immediate memory span, new learning, susceptibility to interference, and recognition memory.
Change From Baseline to Week 8 in the Trail Making Test (TMT-A) | Baseline to Week 8
  TMT-A assesses cognitive processing speed and consists of 25 circles distributed over a sheet of paper. Lower scores represent better speed of processing.
Percentage of participants with MADRS response at week 8 | Baseline to Week 8
  MADRS response was defined as a ≥50% decrease in MADRS total score from baseline
Change from baseline to 8 weeks in the HAM-A (Hamilton Anxiety Rating Scale) | Baseline to Week 8
  HAM-A is a widely used and well-validated tool for measuring the severity of a patient's anxiety, Higher scores indicate greater severity of symptoms.
Change in the quality of life | Baseline to Week 8
  Change from baseline to 8 weeks and endpoint mean scores in FACT-H&N (the Functional Assessment of Cancer Therapy-Head and Neck) Scale，Higher scores indicate greater severity of symptoms.
Change From Baseline to Week 8 in CGI-S (the Clinical Global Impressions-Severity) Score | Baseline to Week 8
  The CGI-S assesses the clinician's impression of the subject's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill).
Dropouts due to adverse events | Baseline to Week 8
  Number of participants who dropped out due to adverse events during the trial
Dropouts due to inefficacy | Baseline to Week 8
  Number of participants who dropped out due to inefficacy during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided